CLINICAL TRIAL: NCT06879951
Title: Evaluation of Serum and Gingival Crevicular Fluid Asprosin Levels in Obese and Normal-Weight Patients with Periodontitis
Brief Title: EVALUATION of GINGIVAL CREVICULAR FLUID and SERUM ASPROSIN LEVELS in OBESE and NORMAL-WEIGHT INDIVIDUALS with PERIODONTITIS
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Collaborators: Gazi University Scientific Research Unit (Unknown)
Responsible Party: Principal Investigator, Buse Naz BÜYÜKAKÇALI ALTAY, Research assistant, Gazi University
Other Study IDs: E-21071282-050.99-720599
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Periodontitis; Obesity
Keywords: Periodontitis; Obesity; Asprosin; Chronic Inflammatory Diseases
MeSH Terms: conditions — Periodontitis; Obesity; Arachnodactyly

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Obese individiuals with periodontitis
  Interventions: Other: Participants are not assigned an intervention as part of the study.
- Obese individuals with periodontal healthy
  Interventions: Other: Participants are not assigned an intervention as part of the study.
- Normal-weight Individuals with Periodontitis
  Interventions: Other: Participants are not assigned an intervention as part of the study.
- Normal-weight Individuals with periodontal health
  Interventions: Other: Participants are not assigned an intervention as part of the study.

INTERVENTIONS:
Other: Participants are not assigned an intervention as part of the study. — Participants are not assigned an intervention as part of the study.

SUMMARY:
Obesity and periodontitis are chronic inflammatory diseases that share common pathological mechanisms. Asprosin, a novel adipokine discovered in 2016, has not been extensively studied in relation to periodontal tissues. In our study, we investigate the levels of asprosin in both serum and gingival crevicular fluid of patients with obesity and those of normal weight who have periodontitis. Additionally, our research aims to clarify the pathophysiological mechanisms linking periodontitis and obesity by examining local and systemic levels of TNF-α, IL-6, and asprosin, alongside clinical periodontal parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to participate in the study.
2. Weight classification:

   * Obese individuals: Body mass index (BMI) of 30 kg/m² or higher.
   * Normal-weight individuals: BMI between 18.5 and 24.9 kg/m².
3. Periodontal health status:

   * Bleeding on probing: less than 10%.
   * Periodontal pocket depth: less than 3 mm.
   * No sites showing attachment loss or alveolar bone loss on radiographs.
4. For individuals with periodontitis:

   * At least two non-adjacent teeth must show signs of interdental attachment loss.
   * Periodontal pocket depth greater than 3 mm.

Exclusion Criteria:

1. Individuals who have received periodontal therapy, any oral decontamination treatment, or antibiotics or steroids in the six months prior to the start of the study.
2. Individuals who are pregnant or breastfeeding.
3. Individuals diagnosed with rheumatoid arthritis or lupus erythematosus.
4. Individuals with a medical history of radiation or cancer therapy.
5. Patients with diabetes, defined by:

   * Hemoglobin A1c (HbA1c) level greater than 6.5%.
   * Fasting blood glucose (FBG) greater than 126 mg/dL.
   * An abnormal oral glucose tolerance test (OGTT).
6. Smokers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients were recruited from the Periodontology Clinic at Gazi University Faculty of Dentistry between August 2023 and August 2024. All participants who met the inclusion criteria were included in the study. Before their participation, the study's purpose and methods were explained, and written informed consent was obtained.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Biyomarker levels | 08.10.2023-08.10.2024
  All groups' GCF and serum levels of asprosin, TNF-α, and IL-6 levels

CONTACTS AND LOCATIONS:
Overall Officials: Aysen Bodur, Professor, Study Director — Gazi University Faculty of Dentistry Department of Periodontology
Locations (1):
- Gazi University Faculty of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No